CLINICAL TRIAL: NCT04812093
Title: Spectroscopic Evaluation of Middle Ear Infection
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Elliot L Botvinick, Professor of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 20163039; R43DC018248 (NIH)
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Middle Ear Infection
Keywords: Middle Ear Infection
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Tool: Spectroscopic otoscope
  Interventions: Device: Spectroscopic otoscope measurements

INTERVENTIONS:
Device: Spectroscopic otoscope measurements — Spectroscopic otoscope measurements are taken with the investigational device. Each measurement consists of placing the device in the ear canal and illuminating the ear with multiple light sources in a short period of time. If wax is present in the ear canal, it is removed by the study physician and another measurement is taken.

SUMMARY:
Otitis media is more common in young children and it is estimated that 75% of all children experience at least one episode before the age of three. Otitis media is one of the common pediatric diagnoses and recurrent episodes account for the most commonly performed surgical procedure. Despite this a high degree of inaccuracy exists in diagnosis of this condition which depends on subjective assessment of the ear drum via direct visualization using an otoscope. Researchers can use LED-based multi wavelength light absorption and scattering measurements for the analysis of ear drum and the middle ear.

DETAILED DESCRIPTION:
The research can use low energy LED signal light sent into the ear canal to measure the tissue optical properties including the absorption of the light signal and the amount of signal that will be backscattered by the tissue components. These measurements will then be analyzed using a microprocessor to determine presence of fluid or inflammation of the eardrum.

ELIGIBILITY:
Inclusion Criteria:

1. Male/ female at all age- newborn to adult.
2. Non- pregnant woman.
3. Diagnose of middle ear infection and plan for surgery procedure.

Exclusion Criteria:

1. Pregnant woman
2. Incompetent adults (i.e. individuals with cognitive impairment)
3. No diagnose of middle ear infection and no plan for surgery procedure.
4. Adults with cognitive impairment and children of parents that are cognitively impaired and thus are unable to consent will be excluded from the study.

Max Age: 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: UCI otolaryngology clinic, CHOC, and La Veta
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Middle Ear Exam | 5 minutes
  The level of light scattering and absorption as measured will be the predictor and presence of fluid behind the ear drum as determined by the surgeon during ear tube placement procedure will be our outcome variable.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Botvinick, Principal Investigator — University of Calfornia Irvine
Locations (2):
- United States (2):
  - Children's Hospital of Orange County (CHOC), Orange, California
  - UCI Otolaryngology Clinic, Orange, California

IPD SHARING:
Plan to Share IPD: No